CLINICAL TRIAL: NCT01443780
Title: Kisel-10- a Prospective Randomized Double-blind Placebo Controlled Study of the Results of Intervention With Selenium and Coenzyme Q10 Combined, Regarding Effect With Emphasis on Cardiovascular Mortality and Morbidity.
Brief Title: Intervention With Selenium and Q10 on Cardiovascular Mortality and Cardiac Function in the Elderly Population in Sweden
Acronym: KiSel-10
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Collaborators: Ostergotland County Council, Sweden (Other); The Swedish Research Council (Other Government); Pharma Nord (Industry)
Responsible Party: Principal Investigator, Urban Alehagen, Principal investigator, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KiSel-10
Record Dates: First submitted 2011-09-28; First posted 2011-09-30 (Estimated); Last update posted 2011-10-03 (Estimated); Status verified 2011-09

CONDITIONS: Cardiovascular Mortality; Cardiac Function
Keywords: Selenium; Q10; dietary supplement; elderly population; intervention; All-cause mortality; cardiac function
MeSH Terms: interventions — Selenium; Tuberculin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- sellenium + Q10 (Experimental): Active dietary supplement that is compared against a placebo arm
  Interventions: Dietary Supplement: Selenium and ubiquinon (Q10) combined
- Sugar pills (Placebo Comparator): Placebo arm that is compared against active intervention with a dietary supplement with selenium + Q10
  Interventions: Dietary Supplement: Selenium and ubiquinon (Q10) combined

INTERVENTIONS:
Dietary Supplement: Selenium and ubiquinon (Q10) combined — A combination of 200 mg/day of coenzyme Q10 (Bio-Quinon 100 mg B.I.D, Pharma Nord, Vejle, Denmark) and 200 µg/day of organic selenium (SelenoPrecise 200 µg, Pharma Nord), or placebo
  Other Names: Bio-Quinon 100mg; SelenoPrecise 200microgr

SUMMARY:
The dietary supplements selenium and Q10 has been evaluated in a double blind placebo-controlled study in an elderly Swedish population. The hypothesis is that as a majority of Northern Europeans suffers insufficient levels of selenium that is used by the cell in the building of at least 25 different enzyme systems in the body, and that the cell need presence of Q10 in order to produce the selenium containing enzymes, we wanted to evaluate the effect of a combined intervention of the two supplements in an elderly population in Sweden. All participants were controlled every 6 months, and the intervention was 48 months in each participant. Besides blood samples, echocardiography and cardiac natriuretic peptides were analyzed at start, every 6 months and at end of the study.

DETAILED DESCRIPTION:
The amount of patients suffering from heart failure is increasing throughout the Western hemisphere. The prognosis of heart failure is poor, in many cases worse than malignant diseases.

Several studies have demonstrated that by evaluating the plasma concentration of the natriuretic peptides that are stimulated by increased wall tension of the myocardium, it is possible to estimate the risk of cardiovascular mortality.

Scientific reports have demonstrated decreased symptoms of heart failure after selenium supplementation. Selenium, which is acquired by the body through food, often exists in low levels in the body in the northern parts of Europe due to poor levels of selenium in the soil. Animal studies have shown that selenium has a positive effect on the myocardium.

Ubiquinon, commonly called Q10, has a central position in many of the enzyme systems of the body. It has recently been shown that the body requires the presence of Q10 to produce selenium containing enzymes which are central in the energy handling processes of cells.

The aim of the present study is to evaluate whether the supplementation of selenium combined with Q10 can influence heart failure and cardiovascular mortality in an elderly population.

In 1998 all people aged between 70-80 years living in the Kinda municipality in Sweden were offered the chance to participate in an epidemiological study with an emphasis on heart failure. Of the 1130 people living in the municipality in the specified age group, 871 agreed to participate in the study. Participants have been questioned regarding a new patient record, examined, new echocardiograms have been performed, blood samples drawn and health related quality of life evaluated. These participants will also be offered the chance to participate in a follow-up of this epidemiological study. In addition to this, they will be offered the chance to participate in the present intervention study where they will be given a dietary supplement of 200 microgram selenium/day and 200 milligram Q10/day, or a placebo.

No serious side effects from these supplements have been observed in earlier studies using the doses planned in this intervention study. The dietary supplements are sold without any restrictions as over the counter products.

During the study all participants will be followed-up with blood samples, a new patient record, and new tablets every six months. Evaluation of health related quality of life will be performed at inclusion, after 18 months and after 48 months. The quality of life will be evaluated using the validated instrument SF-36. At the end of the study, new blood samples and new echocardiograms will be obtained.

Aim To evaluate changes in primarily cardiovascular mortality and all-cause mortality , and secondary, cardiac function as evaluated with cardiac natriuretic peptides and echocardiography after dietary supplementation of selenium and Q10, or a placebo, in an elderly population during 48 months of intervention.

Secondary objectives To evaluate the cost-effectiveness of selenium and Q10 combined during an intervention of 48 months. To measure the perceived health related quality of life during intervention.

Possible health related economic consequences will be evaluated using the instrument EQ-5D.

Endpoint Development of cardiovascular disease, worsening of existing cardiovascular disease, and cardiovascular mortality during intervention with selenium and Q10 in comparison with placebo.

Change of concentration of natriuretic peptides during intervention with selenium and Q10.

Secondary endpoint Development of all-cause mortality during intervention with selenium and Q10. Consumption of hospital resources during intervention with selenium and Q10 in relation to placebo.

Study design A prospective randomized double-blind placebo controlled study. Randomising The randomising procedure will be performed using PharmaNord's computer assisted randomization in blocks of 6.

Study All participants will be offered a selenium-containing yeast preparation corresponding to 200 micrograms of selenium/day, and ubiquinone corresponding to 200 milligrams/day, or a placebo.

During the intervention period, blood samples will be drawn every six months from all participants, and the following list of substances are to be analyzed:

1. NT-proBNP
2. Thioredoxin
3. Thioredoxinreductase
4. Lipidperoxidase
5. Panel of cytokines
6. "New" biomarkers for heart failure. All blood sample results will be blinded for both the investigators and the participants.

Inclusion criteria Individuals living in the municipality of Kinda, aged between 70-80 years who have accepted participation in the study, and who are expected to fulfill a study period of 4 years.

Exclusion criteria Recent myocardial infarction (within 4 weeks). Planned cardio-vascular operative procedure within 4 weeks. Hesitation concerning if the candidate can decide for him/herself whether to participate in the study or not, or if he/she understands the consequences of participation.

Serious disease that substantially reduces survival or where it is not expected that the participant can cooperate for the full 4 year period.

Other factors making participation unreasonable, such as long/complicated transport to the Primary Health Center where the project is managed, or drug/alcohol abuse.

Preparations Coenzyme Q10 ( Bio-Quinon 200mg, PharmaNord, Vejle, Denmark) Selenium (SelenoPrecise 200 microgram, PharmaNord, Vejle, Denmark) Placebo (PharmaNord, Vejle, Denmark) All preparations will be ingested twice a day together with food.

The preparations will be supplied by PharmaNord, Vejle, Denmark. The preparations will be stored in a locked, dry, dark room where only the personnel involved in the study will have access. A rigorous log regarding received and delivered preparations will be kept.

Concomitant pharmacological treatment Participants who have been prescribed pharmacological drugs due to concomitant diseases/medical conditions are advised to continue treatment.

Participants who have been prescribed anticoagulants containing warfarin are advised to continue treatment, but it is recommended that they analyze the INR at the start of the intervention with selenium and Q10, and again after 2 weeks. Interactions between selenium/Q10 and warfarin have been discussed in literature but have not been demonstrated.

Where is the code list? The code list containing information of active treatment/placebo is kept in a sealed envelope at PharmaNord, Vejle, Denmark, and the codes will not be broken before the end of the study, or in the case of an emergency where information regarding the intervention is required.

Side effects Serious side effects should be reported to both the National Board of Health and Welfare and PharmaNord.

Dropouts Participants choosing to discontinue the study for any reason will be followed according to the intention to treat principle. All dropouts will be registered, as well as their reason for discontinuing participation, if the participant chooses to supply this information.

Participants who take supplements of selenium or Q10 for any reason outside the study will be regarded as dropouts.

Ethical permission Ethical permission shall be accepted from the Ethical Review Board before the start of the study. Oral and written "patient" information will be given to all participants, as well as a signed copy of the consent form .

Permission from the Swedish Medical Products Agency Contact has been taken with the Medical Products Agency in Sweden regarding permission to use the preparations during the intervention. However, the principal investigator of the project has been orally informed by the Agency that since this was not regarded as a trial of a medication, but rather of food supplement commodities that are readily available as commercial goods, the Agency would not review the study protocol.

Participants 500-600 healthy individuals as well as patients treated for various diseases and already participating in the former epidemiological heart failure study in the Kinda municipality.

Basic power calculation Using the assumption that the incidence of occurrences in the placebo group during a follow up of 4 years is 40%, and 28% in the intervention group, i.e. a difference in incidence between the groups of 30% and an absolute difference of 12%, 244 individuals are needed in order to obtain a statistical power of 80% with a significance level of 5%. A dropout frequency of 15% is to be expected, which is why a minimum of 560 individuals is needed in order to obtain significant differences.

Principal investigator Urban Alehagen, Resident, Dept of Cardiology, University Hospital of Linköping

Co-investigators Ulf Dahlström, Professor, Dept of Cardiology, University Hospital of Linköping Anders Rosén, Professor, Dept of Cellular Biology, University of Linköping Mikael Björnstedt, Professor, Dept of Pathology, Karolinska University Hospital, Stockholm

ELIGIBILITY:
Inclusion Criteria:

* All elderly persons living in Kinda Municipality,
* Sweden aged 70-87, who have accepted participation in the study, and who are expected to fulfill a study period of 4 years.

Exclusion Criteria:

* Recent myocardial infarction (within 4 weeks).
* Planned cardio-vascular operative procedure within 4 weeks.
* Hesitation concerning if the candidate can decide for him/herself whether to participate in the study or not, or if he/she understands the consequences of participation.
* Serious disease that substantially reduces survival or where it is not expected that the participant can cooperate for the full 4 year period.
* Other factors making participation unreasonable, such as long/complicated transport to the Primary Health Center where the project is managed, or drug/alcohol abuse.

Ages: 70 Years to 87 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 443 (Actual)
Dates: Start 2003-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Change in cardiovascular and all-cause mortality as effect of intervention | From start until 48 months of intervention
  The cardiovascular and all-cause mortality is registered in the study population and an evaluation effect of intervention in terms of change in mortality will be analyzed

SECONDARY OUTCOMES:
Change in cardiac function as measured by echocardiography and cardiac natriuretic peptides as effect of the intervention | From start until 48 months of intervention
  In every participant the cardiac function will be evaluated through echocardiography and cardiac natriuretic peptides. The evaluation through echocardiography will be performed at start and at end of the study, while the cardiac natriuretic peptides will be analyzed every 6 months during the study period. Evaluation of cardiac function will be compared between the two intervention groups (active vs placebo)

CONTACTS AND LOCATIONS:
Overall Officials: Urban Alehagen, PhD, MD, Principal Investigator — Inst of Medicine and Health, University Hospital of Linköping, Sweden
Locations (1):
- Dept of Cardiology, University Hospital of Linköping, Linköping, Sweden

REFERENCES:
- [Derived] Alehagen U, Alexander J, Aaseth JO, Larsson A, Opstad TB. Supplementation with selenium and coenzyme Q10 in an elderly Swedish population low in selenium - positive effects on thyroid hormones, cardiovascular mortality, and quality of life. BMC Med. 2024 May 7;22(1):191. doi: 10.1186/s12916-024-03411-1. PMID 38714999
- [Derived] Alehagen U, Johansson P, Svensson E, Aaseth J, Alexander J. Improved cardiovascular health by supplementation with selenium and coenzyme Q10: applying structural equation modelling (SEM) to clinical outcomes and biomarkers to explore underlying mechanisms in a prospective randomized double-blind placebo-controlled intervention project in Sweden. Eur J Nutr. 2022 Sep;61(6):3135-3148. doi: 10.1007/s00394-022-02876-1. Epub 2022 Apr 6. PMID 35381849
- [Derived] Alehagen U, Aaseth J, Larsson A, Alexander J. Decreased Concentration of Fibroblast Growth Factor 23 (FGF-23) as a Result of Supplementation with Selenium and Coenzyme Q10 in an Elderly Swedish Population: A Sub-Analysis. Cells. 2022 Feb 1;11(3):509. doi: 10.3390/cells11030509. PMID 35159318
- [Derived] Alehagen U, Aaseth J, Alexander J, Johansson P, Larsson A. Supplemental selenium and coenzyme Q10 reduce glycation along with cardiovascular mortality in an elderly population with low selenium status - A four-year, prospective, randomised, double-blind placebo-controlled trial. J Trace Elem Med Biol. 2020 Sep;61:126541. doi: 10.1016/j.jtemb.2020.126541. Epub 2020 May 4. PMID 32417634
- [Derived] Alehagen U, Johansson P, Aaseth J, Alexander J, Surowiec I, Lundstedt-Enkel K, Lundstedt T. Significant Changes in Metabolic Profiles after Intervention with Selenium and Coenzyme Q10 in an Elderly Population. Biomolecules. 2019 Sep 30;9(10):553. doi: 10.3390/biom9100553. PMID 31575091
- [Derived] Alehagen U, Alexander J, Aaseth J, Larsson A. Decrease in inflammatory biomarker concentration by intervention with selenium and coenzyme Q10: a subanalysis of osteopontin, osteoprotergerin, TNFr1, TNFr2 and TWEAK. J Inflamm (Lond). 2019 Mar 18;16:5. doi: 10.1186/s12950-019-0210-6. eCollection 2019. PMID 30923464
- [Derived] Alehagen U, Aaseth J, Alexander J, Johansson P. Still reduced cardiovascular mortality 12 years after supplementation with selenium and coenzyme Q10 for four years: A validation of previous 10-year follow-up results of a prospective randomized double-blind placebo-controlled trial in elderly. PLoS One. 2018 Apr 11;13(4):e0193120. doi: 10.1371/journal.pone.0193120. eCollection 2018. PMID 29641571
- [Derived] Alehagen U, Alexander J, Aaseth J. Supplementation with Selenium and Coenzyme Q10 Reduces Cardiovascular Mortality in Elderly with Low Selenium Status. A Secondary Analysis of a Randomised Clinical Trial. PLoS One. 2016 Jul 1;11(7):e0157541. doi: 10.1371/journal.pone.0157541. eCollection 2016. PMID 27367855
- [Derived] Alehagen U, Johansson P, Bjornstedt M, Rosen A, Dahlstrom U. Cardiovascular mortality and N-terminal-proBNP reduced after combined selenium and coenzyme Q10 supplementation: a 5-year prospective randomized double-blind placebo-controlled trial among elderly Swedish citizens. Int J Cardiol. 2013 Sep 1;167(5):1860-6. doi: 10.1016/j.ijcard.2012.04.156. Epub 2012 May 23. PMID 22626835